CLINICAL TRIAL: NCT01389427
Title: A Multicenter Phase IB Dose Escalation Study to Evaluate the Safety, Feasibility and Efficacy of the Torisel-Rituximab-Cyclophosphamide-Doxorubicin-Vincristine-Prednisone (T-R-CHOP), Torisel-Rituximab-Fludarabine-Cyclophosphamide (T-R-FC) and Torisel-Rituximab-Aracytine High Dose-Dexamethasone (T-R-DHA) for the Treatment of Patients in Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Escalating Doses of Torisel in Combination With Three Chemotherapies Regimens: R-CHOP, R-FC or R-DHA for Patients With Relapsed/Refractory Mantle Cell Lymphoma (MCL).
Acronym: T³
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T³
Record Dates: First submitted 2011-07-04; First posted 2011-07-08 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Mantle Cell Lymphoma Refractory
MeSH Terms: interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Torisel 15 mg (Experimental): Chemotherapy (R-CHOP, R-DHA or R-FC) associated to Torisel 15 mg
  Interventions: Drug: Torisel dose 15 mg and R-CHOP; Drug: Torisel dose 15 mg and R-FC; Drug: Torisel dose 15 mg and R-DHA
- Torisel 25 mg (Experimental): Chemotherapy (R-CHOP, R-DHA or R-FC) associated to Torisel 25 mg
  Interventions: Drug: Torisel dose 25 mg and R-CHOP; Drug: Torisel dose 25 mg and R-FC; Drug: Torisel dose 25 mg and R-DHA
- Torisel 50 mg (Experimental): Chemotherapy (R-CHOP, R-DHA or R-FC) associated to Torisel 50 mg
  Interventions: Drug: Torisel dose 50 mg and R-CHOP; Drug: Torisel dose 50 mg and R-FC; Drug: Torisel dose 50 mg and R-DHA
- Torisel 75 mg (Experimental): Chemotherapy (R-CHOP, R-DHA or R-FC) associated to Torisel 75 mg
  Interventions: Drug: Torisel dose 75 mg and R-CHOP; Drug: Torisel dose 75 mg and R-FC; Drug: Torisel 75 mg and R-DHA

INTERVENTIONS:
Drug: Torisel dose 15 mg and R-CHOP — Torisel in association with Rituximab-Cyclophosphamide-Doxorubicin-Vincristine-Prednisone (R-CHOP) administered every 3 weeks (21 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm A cohort -1
  Arms: Torisel 15 mg
Drug: Torisel dose 15 mg and R-FC — Torisel in association with Rituximab-Fludarabine-Cyclophosphamide (R-FC) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm B cohort -1
  Arms: Torisel 15 mg
Drug: Torisel dose 15 mg and R-DHA — Torisel in association with Rituximab-Aracytine (high dose)-Dexamethasone (R-DHA) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm C cohort -1
  Arms: Torisel 15 mg
Drug: Torisel dose 25 mg and R-CHOP — Torisel in association with Rituximab-Cyclophosphamide-Doxorubicin-Vincristine-Prednisone (R-CHOP) administered every 3 weeks (21 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm A cohort 1
  Arms: Torisel 25 mg
Drug: Torisel dose 50 mg and R-CHOP — Torisel in association with Rituximab-Cyclophosphamide-Doxorubicin-Vincristine-Prednisone (R-CHOP) administered every 3 weeks (21 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm A cohort 2
  Arms: Torisel 50 mg
Drug: Torisel dose 75 mg and R-CHOP — Torisel in association with Rituximab-Cyclophosphamide-Doxorubicin-Vincristine-Prednisone (R-CHOP) administered every 3 weeks (21 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm A cohort 3
  Arms: Torisel 75 mg
Drug: Torisel dose 25 mg and R-FC — Torisel in association with Rituximab-Fludarabine-Cyclophosphamide (R-FC) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm B cohort 1
  Arms: Torisel 25 mg
Drug: Torisel dose 50 mg and R-FC — Torisel in association with Rituximab-Fludarabine-Cyclophosphamide (R-FC) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm B cohort 2
  Arms: Torisel 50 mg
Drug: Torisel dose 75 mg and R-FC — Torisel in association with Rituximab-Fludarabine-Cyclophosphamide (R-FC) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm B cohort 3
  Arms: Torisel 75 mg
Drug: Torisel dose 25 mg and R-DHA — Torisel in association with Rituximab-Aracytine (high dose)-Dexamethasone (R-DHA) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm C cohort 1
  Arms: Torisel 25 mg
Drug: Torisel dose 50 mg and R-DHA — Torisel in association with Rituximab-Aracytine (high dose)-Dexamethasone (R-DHA) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm C cohort 2
  Arms: Torisel 50 mg
Drug: Torisel 75 mg and R-DHA — Torisel in association with Rituximab-Aracytine (high dose)-Dexamethasone (R-DHA) administered every 4 weeks (28 days) for 6 cycles for patients in relapsed/refractory Mantle Cell Lymphoma (MCL).
  Other Names: Arm C cohort 3
  Arms: Torisel 75 mg

SUMMARY:
This is a multicenter, open label, three arms, Phase IB study.

A dose escalation phase of Temsirolimus (Torisel™) administered in intravenous (IV) at day 2, day 8 and day 15 in combination with three chemotherapies regimens for patients in relapsed/refractory Mantle Cell Lymphoma (MCL):

* Rituximab-Cyclophosphamide-Doxorubicin-Vincristine-Prednisone (R-CHOP) administered every 3 weeks for 6 cycles,
* Rituximab-Fludarabine-Cyclophosphamide (R-FC) administered every 4 weeks for 6 cycles,
* Rituximab-Aracytine high dose-Dexamethasone (R-DHA) administered every 4 weeks for 6 cycles.

DETAILED DESCRIPTION:
This is a three arms trial that investigates Temsirolimus (Torisel™) in combination with three chemotherapy regimens (R-CHOP, R-FC or R-DHA).

Primary Objective:

- To assess the feasibility of these three chemotherapy regimens in combination with Temsirolimus (Torisel™) and to assess the incidence of dose limiting toxicities (DLT) during the two first cycles of Temsirolimus (Torisel™) in combination with three chemotherapy regimens in order to determine the maximal tolerate dose (MTD) in a dose escalating study design in a population of patients in relapsed/refractory Mantle Cell Lymphoma (MCL).

Secondary objectives:

* To assess the safety of the association Temsirolimus with the three chemotherapy regimens,
* To determine the efficacy of the association of Temsirolimus (Torisel™) and these three chemotherapy regimens after 4 cycles and after 6 cycles at the end of treatment: response rate and complete response rate (CR), progression-free survival (PFS), response duration (RD) and overall survival (OS).

All subjects who received at least one dose of Temsirolimus (Torisel™) will be considered evaluable and will be included in the safety analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed refractory or relapsed Mantle Cell Lymphoma (at initial diagnosis or relapse),
2. Ann Arbor Stage I-IV with at least one tumor site measurable,
3. Patients who received prior therapy (at least one but no more than three lines therapies) for Mantle Cell Lymphoma (MCL),
4. Aged ≥ 18 years,
5. ECOG performance status 0, 1 or 2,
6. Adequate hepatic and renal function :

   * Serum Glutamic Oxaloacetic Transaminase (SGOT)/AST or Serum Glutamic Pyruvic TransaminaseSGPT/ALT ≤ 3.0 x upper limit of normal (ULN),
   * Serum Total Bilirubin ≤ 1.5 mg/dL (26 μmol/L) except in case of hemolytic anemia,
   * Serum Creatinine ≤ 2 mg/dL (177 μmol/L) or calculated Creatinine Clearance (Cock-croft-Gault formula) of ≥ 50 mL /min
7. Adequate bone marrow reserve :

   * Absolute neutrophil count (ANC) ≥ 1 G/L (1,000 cells/mm³)
   * Platelets count ≥ 50 G/L
   * Hemoglobin ≥ 9.0 g/dL,
8. Signed and date informed consent,
9. Life expectancy of ≥ 90 days (3 months)

Exclusion Criteria:

1. Other types of lymphomas, e.g. B-cell lymphoma,
2. Contraindication to any drug contained in the three chemotherapy regimens (R-CHOP, R-FC, R-DHA),
3. Tested positive for HIV,
4. Active Hepatitis B and/or C,
5. Exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited, to active systemic fungal infection, diagnosis of fever and neutropenia,
6. Any serious active disease or co-morbid medical condition (according to investigator's decision),
7. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form,
8. Received a biological agent for anti-neoplastic intent within 30 days prior to the first dose of study drug,
9. Use of any standard or experimental anti-cancer drug therapy within 30 days prior to the first dose of study drug,
10. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years,
11. Left Ventricular Ejection Fraction < 45% (calculated by echocardiographic or scintigraphic method),
12. Pregnancy or breast feeding women,
13. Women of childbearing potential who not willing to use an adequate method of birth controls for the duration of the study and for twelve months after the end of treatment,
14. Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for twelve months after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | 56 days
  The evaluable for DLT population is the subset of patients from all treated population with a DLT assessment at the two first cycles.

SECONDARY OUTCOMES:
Complete Response Rate(CR) after 4 cycles and at the end of treatment | 28 days up to 42 days after the last treatment dose
  Response at the end of treatment will be assessed after four cycles and at the end of complete treatment if the patient received all planned cycles or at withdrawal. Patients without response assessments (due to whatever reason) will be considered non-responders. A descriptive analysis will also be performed considering as non-responders all patients who relapsed or died during the treatment phase even if they were prematurely withdrawn as responders.
Progression-free survival (PFS) | From the date of inclusion to the date of first documentated disease progression, relapse or death from any cause up to 3 years
  Progression-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse or death from any cause, according to the Cheson 2007 criteria. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
Duration of Response | From the date of first documentation of a response to the date of first documented evidence of progression/relapse or death from any cause up to 3 years
  Duration of response will be measured from the date of first documentation of a response (CR or PR at the end of treatment) to the date of first documented evidence of progression/relapse or death from any cause, according to the Cheson 2007 criteria. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
Overall Response at the end of treatment | 28 days up to 42 days after the last treatment dose
  The same disease response assessment used for complete response rate will be considered to determine the Overall Response Rate. A Patient will be defined as a responder if he/she has a complete response (CR/CRu) or partial response (PR) after four cycles and at the end of treatment. A descriptive analysis will also be performed considering as non-responders all patients who relapsed or died during treatment phase even if they were prematurely withdrawn as responders.
Overall Survival (OS) | From the date of inclusion to the date of first documentated disease progression, relapse or death from any cause up to 3 years
  Overall survival will be measured from the date of inclusion to the date of death from any cause. Patients who are alive at the time of analysis will be censored at the date of the last contact.
Safety of association Temsirolimus with the three chemotherapy regimens | From the date of informed consent signature to 28 days after the last drug administration
  All subjects who received at least one dose of Temsirolimus (Torisel™) will be considered evaluable and will be included in the safety analysis.
  Analysis of safety will be performed by summarizing adverse events, laboratory data, vital signs and ECOG per-formance status. When applicable, a summary of safety data will also be performed by cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Steven LE GOUILL, Professor, Principal Investigator
Locations (11):
- France (11):
  - CHU de Grenoble MICHALLON, Grenoble, Hôpital Nord 217
  - Hôtel Dieu - Université de Nantes, Nantes, Place Alexis Ricordeau
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital Saint Louis, Paris
  - Hôpital Necker, Paris
  - Groupe hospitalier Sud Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Pontchaillou, Rennes
  - CHU de Tours - Hôpital Bretonneau, Tours